CLINICAL TRIAL: NCT06308172
Title: Impact of Single- Versus Double-layer Hysterotomy Closure on Cesarean Niche Development: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSI/2021
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cesarean Section; Dehiscence; Uterine Bleeding; Uterus; Scar; Uterus Abnormal; Cesarean Section Complications
MeSH Terms: conditions — Uterine Hemorrhage; Cicatrix; Uterine Anomalies

STUDY DESIGN:
Masking Description: Patients are recruited and randomly assigned to either the "single-layer" or "double-layer" arm of the study. The randomization process occurs on the day of the cesarean section. Following randomization, patients are informed about their assigned group, and the cesarean section procedure is then carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-layer (Experimental): Patients who are randomized in this arm undergo a single layer-hysterotomy closure
  Interventions: Procedure: Hysterotomy closure
- Double-layer (Experimental): Patients who are randomized in this arm undergo a double layer-hysterotomy closure
  Interventions: Procedure: Hysterotomy closure

INTERVENTIONS:
Procedure: Hysterotomy closure — Hysterotomy closure is done in either one of two ways. Single layer closure consists in a single layer, unlocked suture. Double layer closure consists in a double layer, unlocked suture.

SUMMARY:
The objective of this randomized monocentric study is to assess potential variations in the incidence and severity of isthmocele morbidity among women undergoing cesarean section with either single or double-layer closure of the hysterotomy. Our primary outcome aims to investigate whether there is a reduction in the median duration of intermenstrual spotting in patients belonging to the two respective closure groups

DETAILED DESCRIPTION:
Cesarean section, the most widely performed surgical procedure globally, has seen a significant increase in rates over the past decades, rising from 12.1% in 2000 to 21% in 2015 for various reasons. A recognized complication of cesarean sections is the formation of a uterine niche, commonly referred to as isthmocele. However, the true incidence of this post-operative complication remains uncertain, with reported figures ranging widely from 7% to 80%. The considerable variability in these estimates is attributed in part to the varying sensitivity of diagnostic tools. Moreover, there is a lack of consensus in the literature regarding the definition of a cesarean niche, particularly concerning the dimensions of the defect.

Recent well-designed randomized controlled trials have investigated the long-term outcomes of single versus double-layer hysterotomy closure during C-sections. These studies found no significant differences in isthmocele incidence or intermenstrual spotting. However, limitations such as the lack of correlation between symptom severity and uterine defect dimensions, the inclusion of women in labor, and relatively short follow-up periods are acknowledged weaknesses, prompting the need for further analysis.

Our objective is to compare the outcomes of single versus double-layer hysterotomy closure in terms of intermenstrual spotting and isthmocele incidence in singleton women undergoing elective C-sections. Crucially, standardizing the surgical suturing technique is essential to mitigate potential misleading outcomes resulting from inter-operator variations.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous
* singleton
* age 18-45
* spontaneous pregnancy or autologous assisted fertilization
* gestational age 38-40 weeks
* elective C-section
* informed consent

Exclusion Criteria:

* coagulopathy
* autoimmune diseases
* gestational diabetes
* anticoagulant therapy
* immunosuppressive therapy
* endometriosis
* uterine fibromatosis
* spontaneous labour
* connective tissue diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Intermenstrual bleeding reduction (days) | 6 months
  The primary outcome of the study is to evaluate weather there is a reduction of intermenstrual bleeding in the six months after cesarean section among the two groups of patients.

SECONDARY OUTCOMES:
Intra-operatory time | 6 months
  Evaluate evaluate weather there is a difference in operative time among the two groups of patients
Blood loss | 6 months
  Evaluate any difference in intra-operative blood loss (milliliters of blood)
Analgesics | 6 months
  Evaluate any difference in post-operative use of analgesics
Post-operatory recovery time | 6 months
  Evaluate any difference in post-operative recovery time (days)
Time to full patient mobilization | 6 months
  Evaluate any difference in post-operative time to full mobilization
Isthmocele | 6 months
  Evaluate any difference in isthmocele incidence between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Perugino, MD, Principal Investigator — Ospedale Policlinico Maggiore Ca' Granda Milano
Locations (1):
- Fondazione Cà Granda IRCCS Ospedale Maggiore Policlinico di Milano, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in cesarean section outcomes. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available by may 2025
Access Criteria: Data will be shared upon reasonable request

REFERENCES:
- [Background] Hegde CV. The never ending debate single-layer versus double-layer closure of the uterine incision at cesarean section. J Obstet Gynaecol India. 2014 Aug;64(4):239-40. doi: 10.1007/s13224-014-0573-9. Epub 2014 Jul 23. No abstract available. PMID 25136167
- [Result] Qayum K, Kar I, Sofi J, Panneerselvam H. Single- Versus Double-Layer Uterine Closure After Cesarean Section Delivery: A Systematic Review and Meta-Analysis. Cureus. 2021 Sep 30;13(9):e18405. doi: 10.7759/cureus.18405. eCollection 2021 Sep. PMID 34729282
- [Result] Marchand GJ, Masoud A, King A, Ruther S, Brazil G, Ulibarri H, Parise J, Arroyo A, Coriell C, Goetz S, Christensen A, Sainz K. Effect of single- and double-layer cesarean section closure on residual myometrial thickness and isthmocele - a systematic review and meta-analysis. Turk J Obstet Gynecol. 2021 Dec 24;18(4):322-332. doi: 10.4274/tjod.galenos.2021.71173. PMID 34955322
- [Result] Verberkt C, Stegwee SI, Van der Voet LF, Van Baal WM, Kapiteijn K, Geomini PMAJ, Van Eekelen R, de Groot CJM, de Leeuw RA, Huirne JAF; 2Close study group. Single-layer vs double-layer uterine closure during cesarean delivery: 3-year follow-up of a randomized controlled trial (2Close study). Am J Obstet Gynecol. 2024 Sep;231(3):346.e1-346.e11. doi: 10.1016/j.ajog.2023.12.032. Epub 2023 Dec 26. PMID 38154502
- [Result] Budny-Winska J, Zimmer-Stelmach A, Pomorski M. Impact of selected risk factors on uterine healing after cesarean section in women with single-layer uterine closure: A prospective study using two- and three-dimensional transvaginal ultrasonography. Adv Clin Exp Med. 2022 Jan;31(1):41-48. doi: 10.17219/acem/142519. PMID 34738347
- [Result] Di Spiezio Sardo A, Saccone G, McCurdy R, Bujold E, Bifulco G, Berghella V. Risk of Cesarean scar defect following single- vs double-layer uterine closure: systematic review and meta-analysis of randomized controlled trials. Ultrasound Obstet Gynecol. 2017 Nov;50(5):578-583. doi: 10.1002/uog.17401. Epub 2017 Oct 9. PMID 28070914